CLINICAL TRIAL: NCT02549729
Title: Effect of the Pelvic Floor Training on Pelvic Floor Muscle Strength in Postmenopausal Women With or Without Hormonal Therapy: A Randomized Controlled Trial
Brief Title: Effect of the Pelvic Floor Training in Postmenopausal Women With or Without Hormonal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Flávia Ignácio Antônio Vassimon, PT Master Degree, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.076.422
Record Dates: First submitted 2015-09-01; First posted 2015-09-15 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Weak; Pelvic Floor; Weak; Muscle; Urinary Incontinence
MeSH Terms: conditions — Asthenia; Urinary Incontinence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): Control group not using hormonal replacement therapy will not receive supervised pelvic floor muscle training. This group will be assessed at baseline and up to 12 weeks. For ethics reason at the end of the study women of the control group will be invited to receive the pelvic floor muscle training program. However, this will not be part of the study.
- Exercise (Experimental): Experimental group not using hormonal replacement therapy will receive supervised pelvic floor muscle training.
  Interventions: Behavioral: pelvic floor muscle training
- Hormone Therapy (No Intervention): Experimental group using hormonal replacement therapy will not receive supervised pelvic floor muscle training.
- Exercise and Hormone Therapy (Experimental): Experimental group using hormonal replacement therapy will receive supervised pelvic floor muscle training.
  Interventions: Behavioral: pelvic floor muscle training

INTERVENTIONS:
Behavioral: pelvic floor muscle training — Women will be instructed to perform pelvic floor muscle training daily at home 4 sets of 10 maximum perceived voluntary contraction of the pelvic floor muscle sustained for 6 seconds followed by 5 flick voluntary contraction of the pelvic floor muscle. The 4 sets will be performed in 4 different positions (supine, all four, sit and standing). Twice a week they will receive a supervised session using the same protocol described above.
  Arms: Exercise; Exercise and Hormone Therapy

SUMMARY:
The purpose of this study is to evaluate the effect of pelvic floor muscle training (PFMT) on muscle function of postmenopausal women using or not using hormonal therapy replacement (HTR). The study will evaluate also the prevalence of urinary incontinence reports, its severity and impact on quality of life.

DETAILED DESCRIPTION:
The climacteric period is marked by the decline of estrogens and androgens which represents negative effect on the urogenital system and may present, as a consequence, pelvic floor muscles (PFM) dysfunction and urinary incontinence (UI). The pelvic floor muscles training (PFMT) and hormone therapy (HT) could result in a significant increase in muscle mass with functional improvement and consequent decrease in complaints of urine loss. The aim of this study is to evaluate the effect of PFMT on muscle function, in the presence of UI, severity and impact on quality of life in postmenopausal women with or without HT.

The variable sexual function was abandoned due to the fact that the majority of the women do not presented active sexual life, which is a criteria to answer the questionnaire Index of Female Sexual Function (IFSF), or did not agree to answer the questionnaire. The anxiety scale was also abandoned because it was a tool to assess sexual function in a broader way.

This is a randomized controlled trial. Postmenopausal women will be divided into 4 groups:

* Group 1- without exercise and without HT
* Group 2 - with exercise and without HT
* Group 3 - without exercise and with HT
* Group 4 - with exercise and HT

Women will be evaluated at baseline and up to 12 weeks. The evaluations of the PFM function will be accomplished through the use of vaginal palpation using the Modified Oxford Scale (MOS) and perineometry. The International Consultation on Incontinence Questionnaire- Short Form (ICIQ - SF) will be used to assess reports of UI, quality of life will be evaluated by the SF36 (Medical Outcomes Study 36 - Item Short - Form Health Survey).

The electromyography was not performed because during the collection of data from the pilot sample there was an excess of outcome measures which made the patients' adhesion unfeasible.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with a maximum of ten years of menopause.
* It is considered menopausal cessation of menstrual cycles for more than twelve months (WHO).
* To be included women must have the ability to contract the pelvic floor muscle (PFM) and have never done PFM training.

Exclusion Criteria:

* Women with diabetes mellitus, thyroid disease, hyperprolactinemia, genital prolapse (above grade 1), neuropathy and vasculopathy.
* Those who are intolerant (pain, allergy gel or latex condom or other discomfort) to PFM function evaluation and those that deny answer the questionnaires during the protocol.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Pelvic floor muscle function, evaluated by Perineometry, up to 12 weeks. | Baseline measurement of pelvic floor muscle function, and up to 12 weeks. Control group will be evaluated at baseline and up to 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- School Healthy Center, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Ignacio Antonio F, Herbert RD, Bo K, Rosa-E-Silva ACJS, Lara LAS, Franco MM, Ferreira CHJ. Pelvic floor muscle training increases pelvic floor muscle strength more in post-menopausal women who are not using hormone therapy than in women who are using hormone therapy: a randomised trial. J Physiother. 2018 Jul;64(3):166-171. doi: 10.1016/j.jphys.2018.05.002. Epub 2018 Jun 15. PMID 29914808